CLINICAL TRIAL: NCT07365072
Title: A Randomised Controlled Trial to Evaluate the Impact of Thoracic PRehabilitation With Inspiratory Muscle tRaining cOmpared to Standard prEhabilitation in People With Lung Cancer for Surgical Treatment . The PRIMROSE Trial
Brief Title: The PRIMROSE Trial
Acronym: PRIMROSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea Bay University Health Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRIMROSE
Record Dates: First submitted 2025-09-12; First posted 2026-01-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Lung Resection; Inspiratory Muscle Training; Prehabilitation; Respiratory Complications; Length of Hospital Stay
Keywords: Inspiratory muscle training; Cancer; Lung resection; Prehabilitation; Lung surgery; Randomised control trial; length of hospital stay
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehab plus device (Experimental): Standard Prehab plus inspiratory muscle training device
  Interventions: Device: Inspiratory muscle training (POWERBreathe); Other: Standard Prehab
- Prehab (Active Comparator): Standard Prehab
  Interventions: Other: Standard Prehab

INTERVENTIONS:
Device: Inspiratory muscle training (POWERBreathe) — Resistance training for inspiratory muscles prior to procedure.
  Arms: Prehab plus device
Other: Standard Prehab — Physical optimisation

SUMMARY:
Smoking is a major cause for developing lung cancer. People diagnosed with lung cancer, may be offered surgery which offers a complete cure. Smoking also damages the lungs and compromises a person's lung function, resulting in shortness of breath. Breathlessness limits the ability to carry out daily physical activities and exercise and makes people vulnerable to developing post procedure complications and even death. Some people with surgically treatable lung cancer have a poor ability to exercise and compromised lung function and are not fit for surgery. They will instead be referred for radiation therapy, chemotherapy or palliative care. Surgery is the preferred treatment option.

The pulmonary rehabilitation program (Prehab) improves fitness levels. In addition, it improves the level of breathlessness, exercise capacity and vulnerability of people with lung cancer, with the aim of making them fit for safe surgery. By adding a breathing training device to the Prehab program, the investigators aim to further improve participants fitness for surgery, lower their risk of developing complications and the time spent in hospital after the procedure. The breathing training device is called an inspiratory muscle training device. The hand-held device helps to train and strengthen the breathing muscles, which are then able to work more effectively. After the procedure, participants may be able to breathe and exercise more easily reducing their risk of developing complications and improving outcomes.

The study will compare two groups of people with lung cancer having surgical removal of part of the lung, at a specialist hospital . One group will receive standard Prehab and inspiratory muscle training with the device prior to the procedure; patients in the second group with receive standard Prehab prior to the procedure. Participants will be followed up for twelve months.

DETAILED DESCRIPTION:
To compare inspiratory muscle training (IMT) with standard Prehabilitation (Prehab) to Prehab alone, in people with lung cancer for surgical procedure.

One hundred and thirty-four participants will be recruited for the study (67 for each arm) and with an anticipated attrition rate of 20-25%, one hundred participants will finally be studied.

All adults with lung cancer, aged18 years or over, diagnosed or suspected of non-small cell lung cancer (NSCLC) with surgically resectable disease, who are referred for pre-treatment optimization with Prehab from the lung cancer Multi-Disciplinary Teams (MDTs).

Adults with lung cancer are referred for pre-treatment optimization with Prehab if they meet the following referral criteria: ≥1 Medical Research Council (MRC) dyspnoea score; or ≥1 World Health Organization (WHO) performance status (PS); age ≥ 70 years or frailty index >3; borderline or poor pulmonary function (forced expiratory volume in one second (FEV1) or diffusion capacity for carbon monoxide (DLCO) <50%); sedentary people despite having adequate FEV1 or DLCO. People will be included in the trial if they are capable of giving consent to participation and aged 18 and over.

Additionally, people who have no contraindications to IMT use.

The aim is to evaluate the impact of thoracic Prehab with IMT compared to standard Prehab in reducing post procedural pulmonary complications following surgical resection in people with lung cancer in a randomised control trial.

Descriptive statistics will be used to summarise participants' characteristics and outcome measures. Statistical analyses will be performed using SPSS statistical software, version 20.0 (IBM Corporation, Armonk, NY, USA). Two-sided significance tests will be used (a\0.05). Data will be presented as mean and standard deviation (SD), or median and interquartile range (IQR) for variables with a skewed distribution. Differences between groups in categorical variables will be tested with Chi square or Fisher's exact test. For continuous data the student's t test or the Mann-Whitney U test will be used. The Wilcoxon signed rank test will be used to compare MIP and QoL at T0 and T1 and T2. Relative risk will be calculated for post procedural pulmonary complications (PPCs) graded 1-V using the Clavien Dindo classification and impact of IMT on the study group compared to the control group. Assuming a 36.7 incidence of PPC after the procedure in the control arm and using a significance level of 0.05 and a power of 80%, 50 participants are required in each arm.

ELIGIBILITY:
Inclusion Criteria: Adults with lung cancer with surgically resectable disease who are referred for pre-treatment optimization with Prehab, from the lung cancer Multi-Disciplinary Teams (MDTs).

The referral criteria for Prehab is below:

* ≥1 Medical Research Council (MRC) dyspnoea score
* ≥1 World Health Organization (WHO) performance status (PS)
* Age ≥ 70 years
* Frailty index >3
* Borderline or poor pulmonary function (forced expiratory volume in one second (FEV1) < 50% or diffusion capacity for carbon monoxide (DLCO) <50%)
* Sedentary people despite having adequate FEV1 or DLCO
* People who are eligible for surgical procedures, including endobronchial excision of tumour, or lobectomy, segmental resection, pneumonectomy or wedge resection, either via a minimally invasive approach or a standard thoracotomy approach

Additionally:

* Participants will be included in the trial if they are capable of providing verbal and written consent for Prehab, and written consent for undergoing a surgical procedure for lung cancer
* People over 18 years of age
* All people will be considered regardless of their baseline respiratory muscle strength

Exclusion Criteria: Inclusion criteria not met

* People diagnosed with other cancers namely, metastatic lung cancer, mesothelioma, sarcoma, mediastinal tumours, or benign diseases
* People who decline Prehab
* People who do not consent to Prehab, and do not attend Prehab. People who do not consent to surgery
* People with a high cardiovascular risk for Prehab and awaiting investigations or interventions (including unstable angina and syncope)
* People with a serious concomitant disorder that would compromise safety during Prehab
* People with an abdominal hernia or recent abdominal surgery
* People with a history of spontaneous pneumothorax and/or evidence of large bullae on radiological imaging
* People with an inability to understand written and/or spoken English (only if carers are able to translate)
* People with a perforated ear drum
* People with worsening heart failure signs and symptoms after IMT
* People with pulmonary hypertension
* People who have suffered from or likely to suffer from costochondritis
* If a participant was involved in a similar study, with potential to cause bias or conflict of interest then they will be excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Post procedure complications | On hospital discharge (assessed up to 2 months)
  Post procedure complications following surgical resection in people with lung cancer. This will be graded I-V using the Clavien Dindo Classification. Post procedure complications will be broadly classified as minor (grade 1) and major complications (grade 2-5 where 5 is death). The investigators want to learn from this study, whether an inspiratory muscle trainer helps reduce grade 2 post procedure complications to grade 1 or no complications, and thereby help shorten the length of stay in hospital for people undergoing lung resection surgery. Lower numbers mean a better outcome. Higher numbers mean a worse outcome.

SECONDARY OUTCOMES:
Measure of Quality of Life | At Prehab initial assessment, periprocedural, at hospital discharge (assessed up to 2 months), 1 month post procedure and 3 months post procedure.
  European Organisation for Research and Treatment of Cancer (EORTC) questionnaire (EOTRC QLQ-30). The scores are transformed into a 0-100 range, where 0 is the lowest possible score and 100 is the highest. A higher score indicates a better outcome for functional and global health scores. However, a higher score on the symptom sales represent a greater burden of symptoms and a worse outcome.
Dyspnoea Score | At Prehab initial assessment, every two weeks whilst undergoing Prehab, periprocedural, at hospital discharge (assessed up to 2 months) and 1 month post procedure.
  Medical research council (MRC) dyspnoea score. This scale is measured from 0 to 4. A higher score means worse outcomes. A lower score means better outcomes.
Performance Status | At Prehab initial assessment, every two weeks whilst undergoing Prehab, periprocedural, at hospital discharge (assessed up to 2 months), 1 month post procedure.
  World Health Organization (WHO) performance status. This assigns scores from 0 to 5. A higher score indicates worse outcomes and a lower score indicates better outcomes.
Thoracoscore | At prehab initial assessment and periprocedural.
  The Thoracic Surgery Scoring System is used in thoracic procedures to estimate mortality risk. It calculates risk based on the person co-morbidities and procedure. The Thoracoscore ranges from -7.37 to 7.37. A higher score indicates a potential worse outcome/ more risk. A lower score indicates a potential better outcome/ less risk.
Frailty Index | At Prehab assessment, every two weeks whilst undergoing Prehab, periprocedural, at hospital discharge (assessed up to 2 months) and 1 month post procedure.
  The Clinical Frailty Index is a tool used to assess a persons health status, by measuring the accumulation of health deficits. The scale is 1 to 9. A higher score indicates a greater level frailty and a lower score indicates a lower level of frailty. A higher score is associated with a worse outcome.
Levels of activity | On Prehab initial assessment, every two weeks of Prehab, periprocedural, at hospital discharge (assessed up to 2 months) and 1 month post procedure.
  Categorised as sedentary, lightly active, moderately active and very active.
Maximum Inspiratory Pressure (MIP) | At Prehab initial assessment, periprocedural and at hospital discharge (assessed up to 2 months).
  Measure of respiratory muscle strength. The higher the number the stronger the respiratory muscles are. For healthy adults, normal ranges are 100 to 120cmH20 for men and 70 to 80 cmH20 in women.
Forced expiratory volume in 1 second (FEV1) | At Prehab initial assessment
  The amount of air a person can forcefully exhale in the first second after a deep breath. Ranges are categorized by percentage of predicted range. In normal lung function, 80% or higher is expected. In mild airflow obstruction values ranges vary between 50-79% and severe airflow obstruction ranges between 30-49% and very severe impairment below 30%.
Transfer factor for carbon monoxide (TLCO) | At Prehab initial assessment
  Measures the amount of carbon monoxide (CO) transferred per minute from alveolar gas to red blood cells (RBCs). This is considered normal when 76% to 140% of the predicted value is achieved. Mild, moderate and severe ranges are for values below 76%.
Mortality | At hospital discharge (assessed up to 2 months), 1 month post procedure , 3 months post procedure and 1 year post procedure
  Death rate
Length of hospital admission | On hospital discharge (assessed up to 2 months).
  The numbers of days the participant spent in hospital. A lower number indicates a better outcome. A higher number indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Wakeman, Study Director — Swansea Bay University Health Board
Locations (1):
- Swansea Bay University Health Board, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be confidential and study results will be disseminated collectively on completion

REFERENCES:
- See also: Link to power breathe website - the inspiratory muscle training device to be used as part of the study — https://www.powerbreathe.com/

DOCUMENTS (2):
  • Study Protocol (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT07365072/Prot_000.pdf
  • Informed Consent Form (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT07365072/ICF_001.pdf